CLINICAL TRIAL: NCT04844255
Title: HIV Integrated Personalized Care Approach to the Prevention, Diagnosis, and Control of Salt-sensitive Hypertension: The HIPO CAP DICTSH STUDY
Brief Title: Acute Salt Sensitivity of Blood Pressure
Acronym: AcuteSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mulungushi University (Other)
Collaborators: University of Zambia (Other)
Responsible Party: Principal Investigator, Sepiso K. Masenga, Dr, Mulungushi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PACTR202102852000433
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Blood Pressure
Keywords: salt sensitivity; salt; acute salt sensitivity; Blood pressure; Mean arterial pressure
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Time series design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre and post intervention group (Other): Same individuals are examined before and after taking 2 tablets of salt
  Interventions: Dietary Supplement: dietary salt

INTERVENTIONS:
Dietary Supplement: dietary salt — 2 grams of dietary salt

SUMMARY:
Dietary salt raises blood pressure in certain individuals immediately after ingestion (acute salt sensitivity; ASS) while not affecting others. It is hypothesized that ASS is a risk factor for hypertension. However, no thresholds or diagnostic guideline is available for ASS. This study is the first aim in the main study (HIPO CAP DITSH Study) aimed at determining the threshold or blood pressure cut-offs for ASS upon ingesting dietary salt.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above. Normotensive. If Hypertensive (should be off antihypertensive medication at least 2 weeks prior to the study)

Exclusion Criteria:

* diabetes patients, ill participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Acute salt sensitivity | 160 minutes
  Mean arterial pressure change of 10 mmHg

SECONDARY OUTCOMES:
Diastolic blood pressure change | 160 minutes
  Diastolic blood pressure change of equal to or more than 10 mmHg
Systolic blood pressure change | 160 minutes
  Systolic blood pressure change of equal to or more than 20 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Sepiso K Masenga, PhD, Principal Investigator — Mulungushi University
Locations (1):
- Livingstone Central Hospital, Livingstone, Southern Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available after publication upon request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publishing results
Access Criteria: email and published article (open access)

REFERENCES:
- [Derived] Masenga SK, Hamooya BM, Patel KP, Kirabo A. Erythrocyte glycocalyx sensitivity to sodium is associated with salt sensitivity of blood pressure in women but not men. Front Nutr. 2024 Mar 8;11:1334853. doi: 10.3389/fnut.2024.1334853. eCollection 2024. PMID 38524849